CLINICAL TRIAL: NCT04554212
Title: Blood Flow Restriction Training After Patellar INStability (BRAINS Trial)
Brief Title: Blood Flow Restriction Training After Patellar INStability
Acronym: BRAINS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Caitlin Conley (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Caitlin Conley, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 56541; CDMRP-CDMRP-PR191214 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2020-08-31; First posted 2020-09-18 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Patellar Dislocation; Knee Injuries; Leg Injury; Wounds and Injuries
MeSH Terms: conditions — Patellar Dislocation; Knee Injuries; Leg Injuries; Wounds and Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard Physical Therapy with Sham BFRT (Active Comparator): Participants will undergo 8 weeks of sham blood flow restriction training with cuff inflated to less than 10% occlusion.
  Interventions: Device: Sham Blood Flow Restriction Training
- Standard Physical Therapy with BFRT (Active Comparator): Participants will undergo 8 weeks of blood flow restriction training with cuff inflated to 60% occlusion.
  Interventions: Device: Blood Flow Restriction Training

INTERVENTIONS:
Device: Blood Flow Restriction Training — Participants will undergo 8 weeks of blood flow restriction training with cuff inflated to 60% occlusion.
  Arms: Standard Physical Therapy with BFRT
Device: Sham Blood Flow Restriction Training — Participants will undergo 8 weeks of sham blood flow restriction training with cuff inflated to less than 10% occlusion.
  Arms: Standard Physical Therapy with Sham BFRT

SUMMARY:
This research study is designed to allow health care professionals and researchers to answer many questions about whether a new type of physical therapy called blood flow restriction training (called BFRT) will improve recovery for those with patellar instability.

DETAILED DESCRIPTION:
Participants will randomly be assigned to 1 of 2 groups. This means that neither the participant or their doctor will not choose the treatment, but that the treatment will be randomly selected (like a coin toss). The study treatments is blood flow restriction training (BFRT). BFRT uses an air cuff that is inflated around the top of the thigh. This temporarily limits blood flow to the muscles and may allow the participant to recover strength more quickly after injury. As will be described later, the participant will be closely monitored during all study treatments to make sure they are as safe as possible.

The two groups that participants could be assigned to are:

1. Standard physical therapy
2. Standard physical therapy and BFRT

Physical Therapy Sessions: We are comparing two physical therapy interventions, one is the standard of care and the other is the standard of care plus an additional treatment. Participants have a 50/50 chance of receiving either treatment. If randomized to receive BFRT, the air cuffs will then be placed on the participants' thighs and they will be doing a standardized exercise program that will vary depending on the stage of rehabilitation they are in and as determined by the study personnel. Participants will also complete a standardized course of physical therapy. Activities in physical therapy may include ice over the knee, range of motion exercises to maintain hip strength and gait training exercises as needed.

The following procedures may be performed. Some procedures may not be performed due to time constraints, availability of equipment, and/or by the decision of the investigator. Before initiating physical therapy, participants will be asked some questions including but not limited to the following: age, sex, level of activities, and expectations. Participants will also complete a Sports Activity Scale to determine their physical activity level.

Timeline of Study Visits:

Visit 1 Screening and enrollment: Upon arriving at the clinic or Biomotion Laboratory, potential subjects will have the following assessments: range of motion and knee instability, both of which are the standard of care for a patient with a suspected patellar instability.

After providing informed consent to participate in the study, we will ask you to provide a urine sample and will collect about 2 teaspoons of blood for laboratory testing. The blood will be collected from your arm using standard venipuncture. In addition, we will ask you questions about your medical history including current medications, demographic information, BMI, and smoking status. You will be asked to complete three study questionnaires: the Norwich Patella Instability Score which asks questions about your knee, the Cincinnati Occupational Rating Scale which asks questions about the physical demands of your job or daily life, and a Visual Analogue Scale that will ask you to rate your current pain. You will be randomized to either standard physical therapy or standard physical therapy with BFRT. You have a 50/50 chance of having BFRT. We will also schedule you to go to the BioMotion laboratory for baseline strength testing and to have your first study MRI at the MRISC.

Visit 2 (1 week)

* Knee and Hip Strength
* Walking Biomechanics
* MRI

Visit 3 (5 weeks)

* Knee and Hip Strength
* Questionnaires

Visit 4 (9 weeks)

* Lab specimens collected (urine and about 2 teaspoons of blood)
* Knee and Hip Strength
* Walking Biomechanics
* Questionnaires

Visit 5 (6 months)

* Lab specimens collected (urine and about 2 teaspoons of blood)
* Knee and Hip Strength
* Walking and Running Biomechanics
* Questionnaires

Visit 6 (1 year)

* Lab specimens collected (urine and about 2 teaspoons of blood)
* Knee and Hip Strength
* Walking, Running, and Jumping Biomechanics
* Questionnaires
* MRI

Visit 7 (2 years)

* Lab specimens collected (urine and about 2 teaspoons of blood)
* Knee and Hip Strength
* Walking, Running, and Jumping Biomechanics
* Questionnaires
* MRI

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of traumatic patellar instability (either primary or recurrent) determined by an American Board of Family Medicine certified physician with a Certificate of Added Qualifications in Sports Medicine or licensed Physical Therapist utilizing clinical examination, radiographic imaging, and patients' reports of instability
* Age 14 to 40 years
* Skeletally mature with closed growth plates visualized by radiograph
* A score of 80 or more on the Sports Activity Scale, which corresponds to participating in "running, twisting, turning (tennis, racquetball, handball, ice hockey, field hockey, skiing, wrestling)" at least 1-3 times per week
* Desire to resume pre-injury activity level

Exclusion Criteria:

* Concomitant osteochondral lesion requiring surgical fixation
* Radiographic evidence of osteoarthritis (< Kellgren-Lawrence Grade 2)
* Previous ipsilateral or contralateral knee surgery
* Most recent instability event more than 3 months before enrollment
* History of any inflammatory disorder
* BMI > 35 kg/m2
* Diabetes or uncontrolled hypertension
* Varicose veins or a history of personal or immediate family history (parental or sibling) of deep vein thrombosis
* Pre-existing conditions or previous surgeries that effect the ability to walk
* Planned trips or vacations that will result in the inability to attend 4 consecutive physical therapy sessions

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The Norwich Patellar Instability Scale | Baseline
  The Norwich Patellar Instability (NPI) Scale is a 19-item scale that asks subjects to rate their perceived patellar instability during different tasks, and has been demonstrated to be a valid and responsive tool for assessing patient-reported outcomes for those being treated conservatively or surgically following patellar dislocation. The NPI is scored on a scale of 0 to 100, with lower scores being indicative of less perceived instability
The Norwich Patellar Instability Scale | 5 Weeks
  The Norwich Patellar Instability (NPI) Scale is a 19-item scale that asks subjects to rate their perceived patellar instability during different tasks, and has been demonstrated to be a valid and responsive tool for assessing patient-reported outcomes for those being treated conservatively or surgically following patellar dislocation. The NPI is scored on a scale of 0 to 100, with lower scores being indicative of less perceived instability
The Norwich Patellar Instability Scale | 9 Weeks
  The Norwich Patellar Instability (NPI) Scale is a 19-item scale that asks subjects to rate their perceived patellar instability during different tasks, and has been demonstrated to be a valid and responsive tool for assessing patient-reported outcomes for those being treated conservatively or surgically following patellar dislocation. The NPI is scored on a scale of 0 to 100, with lower scores being indicative of less perceived instability
The Norwich Patellar Instability Scale | 6 Months
  The Norwich Patellar Instability (NPI) Scale is a 19-item scale that asks subjects to rate their perceived patellar instability during different tasks, and has been demonstrated to be a valid and responsive tool for assessing patient-reported outcomes for those being treated conservatively or surgically following patellar dislocation. The NPI is scored on a scale of 0 to 100, with lower scores being indicative of less perceived instability
The Norwich Patellar Instability Scale | 12 Months
  The Norwich Patellar Instability (NPI) Scale is a 19-item scale that asks subjects to rate their perceived patellar instability during different tasks, and has been demonstrated to be a valid and responsive tool for assessing patient-reported outcomes for those being treated conservatively or surgically following patellar dislocation. The NPI is scored on a scale of 0 to 100, with lower scores being indicative of less perceived instability
Quadriceps Strength Symmetry | 1 Week
  Isokinetic Dynamometer will be used. The primary analysis may include the comparison of these observations over multiple time points, with a particular interest in whether there are between-group or within-patient differences.
Quadriceps Strength Symmetry | 5 Weeks
  Isokinetic Dynamometer will be used. The primary analysis may include the comparison of these observations over multiple time points, with a particular interest in whether there are between-group or within-patient differences.
Quadriceps Strength Symmetry | 9 Weeks
  Isokinetic Dynamometer will be used. The primary analysis may include the comparison of these observations over multiple time points, with a particular interest in whether there are between-group or within-patient differences.
Quadriceps Strength Symmetry | 6 Months
  Isokinetic Dynamometer will be used. The primary analysis may include the comparison of these observations over multiple time points, with a particular interest in whether there are between-group or within-patient differences.
Quadriceps Strength Symmetry | 12 Months
  Isokinetic Dynamometer will be used. The primary analysis may include the comparison of these observations over multiple time points, with a particular interest in whether there are between-group or within-patient differences.
MRI T1rho | 1 Week
  Increased T1rho relaxation times have been associated with loss of proteoglycan content. This then corresponds with MRI changes associated with the loss of proteoglycan content. Patients with patellofemoral pain and maltracking have been demonstrated to have significantly greater T1rho relaxation times in the lateral facet of the patella when compared to healthy volunteers.
MRI T1rho | 12 Months
  Increased T1rho relaxation times have been associated with loss of proteoglycan content. This then corresponds with MRI changes associated with the loss of proteoglycan content. Patients with patellofemoral pain and maltracking have been demonstrated to have significantly greater T1rho relaxation times in the lateral facet of the patella when compared to healthy volunteers.

SECONDARY OUTCOMES:
MRI Muscle Volume | 12 Months
  Quadriceps muscle volume (cm2)
The Norwich Patellar Instability Scale | 24 Months
  The Norwich Patellar Instability (NPI) Scale is a 19-item scale that asks subjects to rate their perceived patellar instability during different tasks, and has been demonstrated to be a valid and responsive tool for assessing patient-reported outcomes for those being treated conservatively or surgically following patellar dislocation. The NPI is scored on a scale of 0 to 100, with lower scores being indicative of less perceived instability
Quadriceps Strength Symmetry | 24 Months
  Isokinetic Dynamometer will be used. The primary analysis may include the comparison of these observations over multiple time points, with a particular interest in whether there are between-group or within-patient differences.
MRI Muscle Volume | 24 Months
  Quadriceps muscle volume (cm2)
MRI T1rho | 24 Months
  Increased T1rho relaxation times have been associated with loss of proteoglycan content. This then corresponds with MRI changes associated with the loss of proteoglycan content. Patients with patellofemoral pain and maltracking have been demonstrated to have significantly greater T1rho relaxation times in the lateral facet of the patella when compared to healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Conley, PhD, Study Director — University of Kentucky
Locations (4):
- United States (4):
  - UK Healthcare at Turfland, Lexington, Kentucky
  - University of Kentucky Biomotion Laboratory, Lexington, Kentucky
  - Center for Sports Performance and Research, Foxborough, Massachusetts
  - Foxboro Sports Medicine Clinic, Foxborough, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brightwell BD, Stone A, Li X, Hardy P, Thompson K, Noehren B, Jacobs C. Blood flow Restriction training After patellar INStability (BRAINS Trial). Trials. 2022 Jan 28;23(1):88. doi: 10.1186/s13063-022-06017-1. PMID 35090543